CLINICAL TRIAL: NCT07162623
Title: A Randomized, Double-Blind, Placebo-Controlled, Two-Arms, Prospective, Single-Center Clinical Study to Assess the Safety, Efficacy and In-Use Tolerability of Test Product i.e. Oziva Bioactive Gluta Fizzy in Subjects With Facial Hyperpigmentation
Brief Title: Clinical Study to Assess Safety, Efficacy and In-Use Tolerability of Oziva Bioactive Gluta Fizzy Effervescent Tablets on Subjects With Facial Dark Spots Such as Pimple Marks, Sunspots, Age Spots and Uneven Skin Tone
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NovoBliss Research Pvt Ltd (Other)
Collaborators: Zywie Ventures Pvt Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: NB250030-ZV_1.0_06Aug25
Record Dates: First submitted 2025-08-21; First posted 2025-09-09 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-08

CONDITIONS: Hyperpigmentation
Keywords: dark spots; age spots; pimple spots; uneven skin tone
MeSH Terms: conditions — Hyperpigmentation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oziva Bioactive Gluta Fizzy Effervescent Tablets 4.1 g containing Glutathione (Experimental): Mode of Usage: Dissolve one effervescent tablet in a full glass of water in 200 mL. Allow it to fully dissolve before consuming. For best results, consume the solution immediately after preparation before the fizz ends.
  Frequency: Once Daily Route of administration: Oral Storage Condition: Store at room temperature 15°C to 30°C, away from sunlight
  Interventions: Other: Oziva Bioactive Gluta Fizzy Effervescent Tablets 4.1 g containing Glutathione
- Placebo Effervescent Tablets 4.1 g (Experimental): Mode of Usage: Dissolve one effervescent tablet in a full glass of water in 200 mL. Allow it to fully dissolve before consuming. For best results, consume the solution immediately after preparation before the fizz ends.
  Frequency: Once Daily Route of administration: Oral Storage Condition: Store at room temperature 15°C to 30°C, away from sunlight.
  Interventions: Other: Placebo Effervescent Tablets 4.1 g

INTERVENTIONS:
Other: Oziva Bioactive Gluta Fizzy Effervescent Tablets 4.1 g containing Glutathione — Mode of Usage: Dissolve one effervescent tablet in a full glass of water in 200 mL. Allow it to fully dissolve before consuming. For best results, consume the solution immediately after preparation before the fizz ends.
  Frequency: Once Daily Route of administration: Oral Storage Condition: Store at room temperature 15°C to 30°C, away from sunlight
  Arms: Oziva Bioactive Gluta Fizzy Effervescent Tablets 4.1 g containing Glutathione
Other: Placebo Effervescent Tablets 4.1 g — Mode of Usage: Dissolve one effervescent tablet in a full glass of water in 200 mL. Allow it to fully dissolve before consuming. For best results, consume the solution immediately after preparation before the fizz ends.
  Frequency: Once Daily Route of administration: Oral Storage Condition: Store at room temperature 15°C to 30°C, away from sunlight
  Arms: Placebo Effervescent Tablets 4.1 g

SUMMARY:
This is a randomized, double-blinded, single-centre, two-arms, placebo-controlled, prospective study to evaluate clinical safety, efficacy and in-use tolerability of Test Product i.e. Oziva Bioactive Gluta Fizzy Effervescent tablets in subjects with facial hyperpigmentation and dark spots.

DETAILED DESCRIPTION:
A total of 60 Indian Subjects (30 Subjects per Test Product), including males and non-pregnant, non-lactating females aged between 21 and 55 years (inclusive). Indian Subjects with a Fitzpatrick skin type of III to VI must present with facial hyperpigmentation and dark spots such as tan, pimple marks, sunspots, age spots, uneven skin tone on both side of face at baseline. Participants will be randomized in a 1:1 ratio to received either test Product A or test Product B. the study aims to complete evaluation for 50 Indian Subjects (25 Subjects per Test Product).

The potential subjects will be screened as per the inclusion and exclusion criteria only after obtaining written informed consent from the subjects. Subjects will be contacted telephonically by recruiting department prior to the screening.

There will be total of 3 visits during the study. The duration of the study will be 90 Days (12 weeks) from the enrolment. Subjects will be instructed to visit the facility as per below visits:

* Visit: 01 (Day 01, Week 00): Screening, ICD obtained, Enrolment, Baseline readings.
* Visit 02 (Day 45, Week 06): Product Phase, Evaluations
* Visit 03 (Day 90, Week 12): Evaluations and Product Phase end | End of Study Assessments of Efficacy Parameters before test product(s) usage will be done on Day 01, and after usage of test product(s) on Day 45 (±2 Days) and Day 90(±2 Days)

ELIGIBILITY:
Inclusion Criteria:

* 1) Age: 21 to 55 years (both inclusive) at the time of consent. 2) Sex: Adult male and female having facial hyperpigmentation and dark spots such as tan, pimple marks, sunspots, age spots, uneven skin tone on both side of face.

  3) Females of childbearing potential should have a self-reported negative urine pregnancy test at the time of screening visit.

  4) Subjects with Fitzpatrick Skin Types III to VI, indicating moderate to dark skin tones.

  5) Subjects should not have used any cosmetic, nutraceutical or therapeutic products for skin ageing in last 3 months.

  6) Subjects must be willing to stop using any cosmetics or any medical products for skin ageing for the duration of the study.

  7) Subjects are not allowed to participate in any other study until this study is complete.

  8) Subjects must be willing and able to follow the study directions and to return for all specified visits with the product.

  9) Subjects must agree to record each use of the test products in the subject's diary card on daily basis.

  10) Subjects must agree to record medication use during the study

Exclusion Criteria:

* 1) Subjects who are on steroids for last six months. 2) Subjects who have used any cosmetic, nutraceutical or therapeutic products for skin last three months.

  3) Subjects who are on product which contains kojic acid, glycolic acid, niacinamide, alpha arbutin, Vitamin C and other skin ageing product.

  4) Subjects with other dermatologic diseases whose presence or products could interfere with the assessment of study.

  5) Subjects that are pregnant and/or breastfeeding. 6) The subject has a known allergy or sensitivity to product ingredients. 7) Subjects if do not agree to limit sun exposure to affected areas such as face during prolonged sun exposure.

  8) The subject has any other skin conditions i.e. cuts, scratches, ring worms, etc. which in the opinion of the Investigator, will interfere with the study results or will create undue risk for the subject.

  9) The subject has any of the conditions or factors that the Investigator believes may affect the response of the skin or the interpretation of the test results.

  10) The subject is currently taking or has taken any medication, which the Investigator believes may influence the interpretation of the data.

  11) Any other condition which could warrant exclusion from the study, as per the dermatologist's/investigator's discretion.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Change in skin radiance measured by Glossymeter (Percent) | Baseline (Day 1) to Day 45 (±2 days) and Day 90 (±2 days)
  Comparison of changes within each test product group and between product groups
Change in skin pigmentation and dark spots measured by Mexameter® MX 18 (Percent) | Baseline (Day 1) to Day 45 (±2 days) and Day 90 (±2 days)
  Comparison of changes within each test product group and between product groups

SECONDARY OUTCOMES:
Change in skin elasticity and firmness (R0 and R2 parameters) measured by Cutometer® Dual MPA 580 (Percentage) | Baseline (Day 1) to Day 45 (±2 days) and Day 90 (±2 days)
  Comparison of changes within each test product group and between product groups
Change in skin hydration measured by Corneometer® CM 825 (Percentage) | Baseline (Day 1) to Day 45 (±2 days) and Day 90 (±2 days)
  Comparison of changes within each test product group and between product groups
Change in oxidative stress marker Superoxide Dismutase (SOD) levels (U/mL) | Baseline (Day 1) to Day 90 (±2 days)
  Comparison of changes within each test product group and between product groups
Change in inflammatory markers (C-Reactive Protein and Interleukin-6 [IL-6]) [pg/mL] | Baseline (Day 1) to Day 90 (±2 days)
  Comparison of changes within each test product group and between product groups
Change in skin color parameters (L*, a*, b*, and ITA) measured by Skin Colorimeter CL 400 (values; ITA in degrees) | Baseline (Day 1) to Day 45 (±2 days) and Day 90 (±2 days)
  Comparison of changes within each test product group and between product groups.
Change in spot color intensity, average size (mm2) and number, pigmentation intensity, and contrast measured by Dermatological Evaluation using Modified Griffiths 10-point Scale | Baseline (Day 1) to Day 45 (±2 days) and Day 90 (±2 days)
  Comparison of changes within each test product group and between product groups
Change in pigmentation intensity, spot surface area (mm2), and skin radiance measured by Image-Pro Analysis | Baseline (Day 1) to Day 45 (±2 days) and Day 90 (±2 days)
  Comparison of changes within each test product group and between product groups
Change in melasma severity measured by Dermatological Evaluation using Melasma Area and Severity Index (MASI) (percentage) | Baseline (Day 1) to Day 45 (±2 days) and Day 90 (±2 days)
  Comparison of changes within each test product group and between product groups
Change in visual skin appearance from facial photographs using Nikon Digital Camera D3300 or equivalent | Baseline (Day 1) to Day 45 (±2 days) and Day 90 (±2 days)
  Comparison of changes within each test product group and between product groups
Change in subject-reported product perception (skin appearance, radiance, pigment reduction, glow, blemishes, and dark patch reduction) assessed by questionnaire | Baseline (Day 1) to Day 45 (±2 days) and Day 90 (±2 days)
  Comparison of responses within each test product group and between product groups

CONTACTS AND LOCATIONS:
Overall Officials: Nayan Patel, Principal Investigator — NovoBliss Research Pvt Ltd
Locations (1):
- NovoBliss Research Private Limited, Ahmedabad, Gujarat, India

IPD SHARING:
Plan to Share IPD: No